CLINICAL TRIAL: NCT02241733
Title: Sustainability of Rehabilitation Gains in COPD
Brief Title: Sustainability of Pulmonary Rehab Gains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: O1325-R
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: COPD
Keywords: exercise; pulmonary rehabilitation; dynamic hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise (Active Comparator): Patients will exercise for 12 weeks and then participate in an adherence program
  Interventions: Behavioral: Exercise only
- exercise plus breathing retraining (Experimental): Patients will exercise plus breathing retraining for 12 weeks and then participate in an adherence program
  Interventions: Behavioral: Breathing retraining plus exercise

INTERVENTIONS:
Behavioral: Breathing retraining plus exercise — Patients will participate in a 12-week exercise program with breathing retraining. They will also participate in an adherence program.
  Arms: exercise plus breathing retraining
Behavioral: Exercise only — Patients will participate in a 12-week exercise program . They will also participate in an adherence program.
  Arms: exercise

SUMMARY:
People with moderate to severe COPD trap air in their lungs. This lessens their ability to exercise. The investigators developed a computerized breathing retraining program to help patients empty their lungs during exercise. The investigators believe that learning to control breathing will help patients be more active. The purpose of this study is to test the effects of using breathing retraining (intervention group) versus no breathing retraining (control group) as part of a 12-week exercise program. The investigators are examining the long term effects of this training on exercise capacity and the ability to empty ones lungs during exercise. Patients will participate in a 12-week exercise program, with or without breathing retraining. They will then participate in a 42 week adherence program to maintain physical activity. Patient testing will be competed at baseline, 12 weeks, 6 months and 1 year. 250 patients with moderate to severe COPD will be enrolled.

DETAILED DESCRIPTION:
Rationale: Development of dynamic hyperinflation is a primary limiting factor of exercise tolerance in chronic obstructive pulmonary disease (COPD). To lessen the development of dynamic hyperinflation, and to improve exercise tolerance in COPD patients, the investigators have developed a breathing-retraining technique to be used during pulmonary rehabilitation. This breathing-retraining technique is designed to decrease respiratory rate and prolong exhalation. The investigators demonstrated that, in the short-term, hyperinflation and exercise duration improved more with breathing-retraining plus exercise-training than with exercise-training alone. Because a crucial aspect of pulmonary rehabilitation is the maintenance its short-term benefits over the long-term, the investigators now propose to test whether short-term benefits of breathing-retraining plus exercise followed by an adherence-intervention program are sustainable over the long-term Primary Hypothesis: (H1) In COPD patients, improvements in exercise duration on a constant- load treadmill test will be greater after 12 weeks of breathing-retraining plus exercise-training followed by a 42-week adherence-intervention program (1 yr. total) than after 12 weeks of exercise-training alone followed by a 42-week adherence-intervention program (1 yr. total). Secondary Hypotheses: One year after randomization, exercise-induced dynamic hyperinflation will be less during a constant-load treadmill test (H2), 6-minute walking distance will be longer (H3), and mastery over breathing will be greater (H4) in the breathing-retraining plus exercise-training group than in the exercise-alone group. Lastly (exploratory objective), the investigators will assess the effect of the patient's physiologic, psychologic and clinical phenotype on short- term and long-term responsiveness to pulmonary rehabilitation.

Methods: The proposed study is a randomized, controlled clinical trial in which 250 patients with moderate-to-severe COPD will be enrolled. One hundred forty of these patients are expected to qualify for randomization into the breathing-retraining plus exercise-training group or the exercise-training alone group. Patients will receive 12-weeks of supervised training according to group assignment (three times weekly) followed by an adherence-intervention program (weekly phone motivational interviews, home-exercise program, and monthly laboratory booster sessions). Follow-up testing will be completed at 12 weeks, and at 6 and 12 months. Testing will include pulmonary function test, incremental-load and constant-load treadmill tests, 6-minute walk test, measurements of dyspnea, assessment of respiratory and quadriceps muscle strength and endurance and quadriceps ultrasonography. Analysis: In the principal analysis of the primary outcome measure (exercise duration; H1) the investigators will compare changes in exercise duration (constant work-rate treadmill test) from baseline to end of study using 2-sample t-test (two-tailed =.05). The primary analysis will be based on intention-to-treat principles. Multiple imputation will be used for study subjects missing the 12-month measurement. This imputation model will be based on baseline characteristics of study participants. Several secondary analyses of the primary outcome measure will be performed (H2-H4). Linear regression will be used to determine whether the observed treatment benefits persist after adjustment for baseline covariates and measures of adherence to treatment. Since several measurements will be taken on each patient, mixed-models analysis will be used to compare the changes on the constant-load treadmill test over time between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* >/= 40 yrs
* FEV1 </= 70% predicted
* FEV1/FVC <70% predicted
* RV/TLC >/=120%
* SpO2 >/= 90% at peak exercise (with or without exercise)
* inspiratory capacity decline >.15L from rest to peak exercise

Exclusion Criteria:

* respiratory infection/exacerbation within the previous 4 weeks
* exercise limiting heart disease
* primary asthma
* congestive heart failure
* exercise limiting peripheral arterial disease
* stops exercise due to arthritic pain in the knee or hips
* inability to walk on the treadmill
* pregnancy
* methadone use
* any unforeseen illness or disability that would preclude exercise testing or training
* participation in a formal exercise program within the previous 12 weeks

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-10-21 (Actual); Study Completion 2019-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen G. Collins, PhD RN, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise: Patients exercised for 12 weeks and then participated in an adherence program
  Exercise only: Patients participated in a 12-week exercise program . They also participated in an adherence program.
- Exercise Plus Breathing Retraining: Patients exercised plus received breathing retraining for 12 weeks and then participated in an adherence program
  Breathing retraining plus exercise: Patients participated in a 12-week exercise program with breathing retraining. They also participated in an adherence program.
Period: Overall Study
Arm/Group | Exercise | Exercise Plus Breathing Retraining
Started | 40 | 40
Completed | 25 | 30
Not Completed | 15 | 10
Not completed — Lost to Follow-up | 9 | 4
Not completed — Physician Decision | 6 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | Exercise Plus Breathing Retraining | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (6.6) | 68.3 (6.6) | 67.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 38 | 39 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 36 | 39 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 29 | 32 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80
Time walked on constant workload treadmill test [Mean (Standard Deviation); unit: minutes walked] | 7.2 (1.9) | 7.1 (2.0) | 7.2 (1.9)
Inspiratory capacity [Mean (Standard Deviation); unit: liters] | 2.09 (.69) | 1.88 (.49) | 1.99 (.59)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Exercise Time on a Constant Work-rate Treadmill Test
Description: Patients walk on a treadmill set at a constant workrate. The difference in the time walked on the treadmill from baseline to study completion is the primary outcome measure.
Time Frame: 52 week test
Population: A multiple imputation model was used to impute missing values for those who did not complete the 52 weeks of the program.
Measure: Mean (Standard Deviation); unit: change in number of minutes walked
Arm/Group | Exercise | Exercise Plus Breathing Retraining
Number analyzed (Participants) | 40 | 40
change in number of minutes walked | 12.2 (3.5) | 12.5 (3.5)
Statistical Analysis 1: Comparison: Exercise vs Exercise Plus Breathing Retraining; An independent t-test was completed; Test type: Superiority; p = 0.94, t-test, 2 sided

2. Secondary Outcome: Inspiratory Capacity
Description: Inspiratory capacity is measured at a set time during the constant workrate treadmill test. The difference between the inspiratory capacity measured at baseline and 52 weeks is a secondary outcome. Inspiratory capacity measured during exercise is a measure of dynamic hyperinflation.
Time Frame: 52 week test
Population: A multiple imputation model was used to impute values for those who did not complete the program. The score below is the difference between 52 weeks and baseline.
Measure: Mean (Standard Deviation); unit: difference in liters inspired
Arm/Group | Exercise | Exercise Plus Breathing Retraining
Number analyzed (Participants) | 40 | 40
difference in liters inspired | -0.02 (.07) | .15 (.07)
Statistical Analysis 1: Comparison: Exercise vs Exercise Plus Breathing Retraining; Test type: Superiority; p = 0.078, t-test, 2 sided

3. Secondary Outcome: 6 Minute Walk Distance
Description: Six-minute walk distance will be measured at 52 weeks. The difference in distance walked in meters between baseline and 52 weeks is the secondary outcome measure. The 6 minute walk is conducted using the guidelines issued by the American Thoracic Society.
Time Frame: 52 weeks
Population: Multiple imputation procedures were used to impute data for those that did not complete the protocol
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Exercise | Exercise Plus Breathing Retraining
Number analyzed (Participants) | 40 | 40
meters | 25.9 (8.5) | 22.8 (8.7)
Statistical Analysis 1: Comparison: Exercise vs Exercise Plus Breathing Retraining; Test type: Superiority; p = 0.80, t-test, 2 sided

4. Secondary Outcome: Mastery Over Breathing
Description: Mastery over breathing is measured using the Chronic Respiratory Disease Questionnaire. Specifically the subscale 'mastery" is the investigators' secondary outcome. The difference in scores from baseline to 52 weeks is the investigators' outcome measure. The Chronic Respiratory Disease Questionnaire is a valid and reliable questionnaire. 1=minimum score, 7=maximum with the higher score indicating greater mastery. A higher score indicates better health. A change of 0.5 indicates a small change, 1.0 indicates a moderate change and greater or equal to a change of 1.5 indicates a large change.
Time Frame: 52 weeks
Population: Multiple imputation was used to impute missing values for those who did not complete the protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise | Exercise Plus Breathing Retraining
Number analyzed (Participants) | 40 | 40
score on a scale | 1.9 (4.9) | 2.3 (4.6)
Statistical Analysis 1: Comparison: Exercise vs Exercise Plus Breathing Retraining; Test type: Superiority; p = 0.76, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of study participation (1 year or the time the patients remained in the study).
Arm/Group | Exercise | Exercise Plus Breathing Retraining
All-Cause Mortality (participants affected / at risk) | 1/40 | 2/40
Serious Adverse Events (participants affected / at risk) | 16/40 | 15/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise (N=40) | Exercise Plus Breathing Retraining (N=40)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 11 (11) — Exacerbation requiring hospitalization or ED visit
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Atrial fibrillation with rapid ventricular response. Required hospitalization.
Rectal abscess (Gastrointestinal disorders) | 1 (1) | 0 (0) — Hospitalized for severe rectal abscess
Kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0) — hospitalized for kidney stones
brain aneurysm (Nervous system disorders) | 1 (1) | 0 (0) — patient hospitalized and died from brain aneurysm
cellulitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Patient developed severe cellulitis of the leg and was hospitalized
meningioma (Nervous system disorders) | 0 (0) | 1 (1)
leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — patient developed leukemia and died
stroke (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT02241733/Prot_SAP_000.pdf